CLINICAL TRIAL: NCT04384198
Title: TransCranial Doppler for REDUCtion of Silent strokE During MitraClip Implantation
Acronym: TCD-REDUCE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Berlin Institute of Health (Other)
Responsible Party: Principal Investigator, Christian Nolte, Prof. Dr. Christian H. Nolte, Charite University, Berlin, Germany
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: EA4/193/19
Record Dates: First submitted 2020-04-30; First posted 2020-05-12 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Mitral Valve Insufficiency
Keywords: MitraClip; Sonolysis; Stroke
MeSH Terms: conditions — Mitral Valve Insufficiency; Stroke

STUDY DESIGN:
Intervention Model Description: PROBE
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sonolysis group (Experimental): Cerebral hemisphere with sonolysis during MitraClip implantation.
  Interventions: Procedure: Sonolysis
- Control group (No Intervention): Cerebral hemisphere without sonolysis during MitraClip implantation.

INTERVENTIONS:
Procedure: Sonolysis — Continuous transcranial Doppler sonography (TCD) using a 2-MHz diagnostic probe with maximal diagnostic energy
  Arms: Sonolysis group

SUMMARY:
The primary goal of the TCD-REDUCE study is to demonstrate the effectiveness of continuous transcranial Doppler sonography ("sonolysis") on the reduction of the ischemic stroke volume during MitraClip implantation.

DETAILED DESCRIPTION:
Cardiac procedures are associated with new cerebral ischemic lesions detected on diffusion-weighted MRI (Bendszus et al., 2006).

A previous study suggests that sonolysis (continuous transcranial Doppler sonography using a 2-MHz diagnostic probe) can reduce the risk of new cerebral ischemic lesions during carotid endarterectomy and carotid angioplasty / stenting (Skoloudik et al., 2015).

Currently, it is unknown whether sonolysis can also reduce the risk of new cerebral ischemic lesions during MitraClip implantation - a percutaneous treatment option in patients with moderate / severe mitral regurgitation.

In this study, patients will receive cerebral MRI and clinical neurological / neuropsychological examination before and after MitraClip implantation. During MitraClip implantation, all patients will receive continuous transcranial Doppler sonography using a 2-MHz diagnostic probe with maximal diagnostic energy administered through either the left or the right transtemporal window (computer-generated 1:1 randomization).

The primary endpoint is the median ischemic lesion volume detected on diffusion-weighted MRI after MitraClip implantation in the sonolysis group and in the control group.

ELIGIBILITY:
Inclusion Criteria:

Patients with mitral regurgitation that are assigned to the MitraClip implantation by an interdisciplinary heart team according to current guidelines.

Exclusion Criteria:

* contraindication to MRI examination (e.g. pace-maker, implanted metal material, claustrophobia)
* pregnancy
* unable to consent
* no transtemporal window

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2020-08-13 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
stroke volume | 0-5 days after the MitraClip Implantation
  median volume (in ml) of new ischemic lesions detected on diffusion-weighted MRI after MitraClip implantation in the sonolysis and in the control group

SECONDARY OUTCOMES:
diffusion-weighted MRI lesions | 0-5 days after the MitraClip Implantation
  new ischemic lesions (occurrence, number and location) detected on diffusion-weighted MRI after MitraClip implantation
intracerebral hemorrhage (ICH) and / or subarachnoid hemorrhage (SAH) | 0-5 days after the MitraClip Implantation
  new ICH and / or SAH detected on T2*-weighted MRI after MitraClip implantation
cerebral microbleeds (CMB) | 0-5 days after the MitraClip Implantation
  new cerebral microbleeds detected on T2*-weighted MRI after MitraClip implantation (occurrence, number and location)
clinically overt stroke | (1) 0-5 days after the MitraClip Implantation and (2) 3 months after MitraClip implantation
  new clinically overt stroke (ischemic or hemorrhagic) or transient ischemic attack (TIA) after MitraClip implantation
functional outcome | (1) 0-5 days after the MitraClip Implantation and (2) 3 months after MitraClip implantation
  functional outcome will be evaluated using the modified Rankin scale (mRS). The mRS ranges from 0 to 6 with 0 indicating no functional deficit (best score) and 6 indicating deaths (worst score).
cognitive outcome during hospital stay | 0-5 days after the MitraClip Implantation
  cognitive outcome will be evaluated using the Montreal Cognitive Assessment (MoCA)
cognitive outcome at follow-up | 3 months after MitraClip implantation
  cognitive outcome will be evaluated using the Telephone Interview for Cognitive Status (TICS)
delirium | 0-5 days after the MitraClip Implantation
  delirium will be evaluated using the 3-Minute Diagnostic Interview for Confusion Assessment Method (3D-CAM)
length of hospital stay (duration of hospitalization for the MitraClip implantation) | length of hospital stay (up to 3 months after MitraClip implantation)
  days of hospital stay from admission to hospital to discharge from hospital including direction of discharge (home, another hospital)
mortality | up to 3 months after MitraClip implantation
  mortality

CONTACTS AND LOCATIONS:
Overall Officials: Christian H Nolte, Prof., Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité-Campus Benjamin Franklin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Skoloudik D, Kuliha M, Hrbac T, Jonszta T, Herzig R; SONOBUSTER Trial Group. Sonolysis in Prevention of Brain Infarction During Carotid Endarterectomy and Stenting (SONOBUSTER): a randomized, controlled trial. Eur Heart J. 2016 Oct 21;37(40):3096-3102. doi: 10.1093/eurheartj/ehv492. Epub 2015 Sep 28. PMID 26417059